CLINICAL TRIAL: NCT06178822
Title: Towards Novel BIOmarkers to Diagnose SEPsis on the Emergency Room
Acronym: BIOSEP
Status: Recruiting | Type: Observational
Sponsor: Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Flevoziekenhuis (Other)
Responsible Party: Principal Investigator, W. J. Wiersinga, MD, Prof. dr. W.J. Wiersinga, MD, Amsterdam UMC, location AMC
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: BIOSEP
Record Dates: First submitted 2023-11-23; First posted 2023-12-21 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-02

CONDITIONS: Sepsis; Septic Shock; Sepsis, Severe; Infections; Infection Viral; Infection, Bacterial; Infections, Respiratory
Keywords: Biomarkers; Emergency Room; A&E; Accident & Emergency
MeSH Terms: conditions — Sepsis; Shock, Septic; Infections; Virus Diseases; Bacterial Infections; Respiratory Tract Infections; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood samples (EDTA, heparin, PaxGene) and rectal swabs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with infection: Patients with an (suspected) infection and a MEWS score 2 or higher
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention

SUMMARY:
Objectives:

1. To compare the immune response of patients with or without sepsis presenting to the ED with a(n) (suspected) infection.
2. To determine immune response aberrations that are associated with an increased risk of developing sepsis in patients presenting to the ED with a(n) (suspected) infection without sepsis.
3. To determine the long term cognitive and physical sequelae of sepsis after admission.

DETAILED DESCRIPTION:
Sepsis will be defined in accordance with the current Sepsis 3.0 criteria as a(n) (suspected) infection with evidence of organ failure, as reflected by a SOFA (Sequential Organ Failure Assessment) score of ≥2. Notably, a molecular definition of sepsis does not exist and there is no pathological gold standard; therefore, in accordance with the current international consensus, the investigators consider the commonly used clinical organ failure (SOFA) criteria as the best option. The SOFA score is composed of six organ dysfunctions (cardiovascular, pulmonary, renal, hepatic, coagulation and neurological). The SOFA score was developed for ICU patients, but its components can be easily scored in an ED (and hospital ward) setting with the exception of the pulmonary component; this pulmonary dysfunction score is based on the PaO2/FiO2 (PF) ratio, wherein PaO2 is the partial pressure of oxygen in arterial blood and FiO2 the fraction of inspired oxygen. Measurement of the PaO2 requires an arterial blood puncture, which is not routinely done on the ER or hospital ward. Therefore, the investigators will use an alternative method to determine the respiratory SOFA by determining the SpO2/FiO2 (SF) ratio, wherein SpO2 is peripheral oxygen saturation. SpO2 is routinely measured by finger pulse oximeter in patients with suspected infection; FiO2 is 21% when breathing room temperature and increases by 4% with each liter of oxygen provided per minute to a patient via a nasal cannula. Cut-off values for SF ratios correlating with SOFA pulmonary scores based on PF ratios have been validated in large data sets.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or higher
* Presentation at the Emergency Department (ED)
* Clinical suspicion of infection or earlier confirmed infection
* Modified Early Warning Score (MEWS) of 2 or higher

Exclusion Criteria:

* No informed consent given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research population will include adult patients that present to the ED of participating hospitals. In order to be eligible to participate in the BIOSEP study there must also be a clinical suspicion of an infection or a confirmed infection and MEWS of 2 or higher.
Sampling Method: Non-Probability Sample
Enrollment: 3300 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Final diagnosis for hospitalization | 4 years
  Adjudicated diagnoses for hospitalization
Disease severity | During hospitalization (up to day 180)
  Sequential Organ Failure Assesment (SOFA) score (minimum 0, maximum 24) collected during admission
Mortality | 4 years
  Mortality at day 30

SECONDARY OUTCOMES:
Length of stay | During hospitalization (up to day 180)
  Both hospital and ICU stay
Mortality | 5 years
  Hospital, ICU, 28-day, 90-day and 1 year mortality
Post-sepsis sequelae | Up to 1 year after sepsis episode
  Up to 1 year post sepsis, e.g. decreased executive functions, weakness, fatigue etc.)
Readmissions | 5 years
  All cause readmissions in the first year after discharge

OTHER OUTCOMES:
Site of infection | 4 years
  Site of infection
Initiated therapies during admission | 4 years
  Initiated therapies during admission

CONTACTS AND LOCATIONS:
Overall Officials: Willem Joost Wiersinga, MD, PhD, Principal Investigator — Amsterdam UMC, location AMC
Locations (3):
- Netherlands (3):
  - Flevoziekenhuis, Almere Stad, Flevoland
  - Amsterdam UMC, location VUMC, Amsterdam, North Holland
  - Amsterdam UMC, location AMC, Amsterdam, North Holland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Reijnders E, Turgman O, Joosten SCM, Schinkel M, Slim MA, Douma RA, Moeniralam HS, Peters-Sengers H, van der Poll T, Wiersinga WJ. Towards novel BIOmarkers to diagnose SEPsis (BIOSEP) in the emergency room: a protocol for a multicentre, prospective cohort study. BMJ Open. 2025 Aug 1;15(7):e103138. doi: 10.1136/bmjopen-2025-103138. PMID 40750284